CLINICAL TRIAL: NCT04790357
Title: Assessment of One-shot Cardiac-cervical-intracranial MRI in the Etiological Work up of Ischemic Stroke and Transient Ischemic Attacks
Acronym: Concise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0394; 2020-A00071-38 (Other: IDRCB)
Record Dates: First submitted 2020-04-10; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference strategy (Other): correspond to the reference techniques according to the current guidelines in the etiological work up of ischemic strokes and TIA
  Interventions: Other: Current guidelines
- Evaluated strategy (Other): correspond to perform the cci-MR: cardiac MRI with late-enhancement, angio-MRI of the cervical and intracranial arteries
  Interventions: Other: cc-MRI

INTERVENTIONS:
Other: Current guidelines — doppler ultrasound and/or angio CT-scan of the cervical arteries, angio CT-scan of the intracranial arteries, TTE wich can be supplemented by a TEE at the discretion of the investigator. The TEE is not mandatory
  Arms: Reference strategy
Other: cc-MRI — of one-shot cardiac-cervical-intracranial MRI: cardiac MRI with late-enhancement, angio-MRI of the cervical and intracranial arteries
  Arms: Evaluated strategy

SUMMARY:
Stroke is a major public health issue in developed countries. A full etiological work up within a short time is critical to implement the appropriate preventive treatment. The etiological work up is actually based on a clinical examination and on a group of paraclinical examinations. The realization of the standard strategy is time consuming, and increase the cost of the medical care. A non-invasive one-shot examination of the heart, the aorta and the cervical and intracranial arteries (cci-MRI) could overcome these disadvantages.The investigator therefore propose to carry out an overall assessment of the performance of the cci-MR in the etiological work up of ischemic strokes and TIAs compared to the reference strategy

ELIGIBILITY:
Inclusion Criteria:

* • Man or woman aged from 18 to 85 years old,
* Patients victims of an ischemic stroke or a TIA in the 2 days before inclusion, Symptoms thought to be consistent with TIA were those defined by the ad hoc Committee established by the Advisory Council for the National Institute of Neurological and Communicative Disorders and Stroke65
* Rankin score: mRS ≤3
* Patient having given their free written and informed consent, or preliminary oral informed consent attested by a third party followed by signed informed consent as soon as possible,
* Affiliated to a social security scheme or equivalent,
* That are not the subject of any legal protection measures

Exclusion Criteria:

* •TIA symptoms limited to isolated numbness,
* changes, or isolated dizziness/vertigo
* Agitation, severe swallowing
* Contraindication to an MRI and the injection of gadolinium,
* Known history of hypersensitivity to the MRI contrast product,
* Risk of pregnancy or known pregnancy revealed when questioned, Breastfeeding,
* Patient unable to understand or poorly understanding French.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the consistency between the reference strategy and the cci-MR strategy for etiological work up according to the ASCOD classification, in ischemic stroke and TIA patients | Within 8 days after hospitalization
  The primary endpoint will be based on the consistency for each patient of the etiological work up according to the ASCOD classification evaluated with cci-MR in comparison of the reference strategy

SECONDARY OUTCOMES:
To assess the reproducibility of the assessment of the cci-MR results | Within 8 days after hospitalization
  The reproducibility of the assessment of the cci-MR results will be based on the following endpoints:
  - Double reading; Concordance intra and inter reviewer
To evaluate the agreement between cci-MR and the reference method for each etiological subgroup: in the context of ischemic stroke or TIA. | Within 8 days after hospitalization
  Agreement for each etiological subgroup between cci-MR and the reference method.
To assess the improvement of the detection of myocardial scar with cci-MR compared to reference strategy | Within 8 days after hospitalization
  Presence or absence of ischemic myocardial scar
To assess the atherosclerotic burden (coronary, intracranial, cervical, aortic) assessed with cci-MR compared to the reference strategy, | Within 8 days after hospitalization
  Presence or absence of coronary, intracranial, cervical, aortic atheroma. The diagnostic work up will focus on cervical artery stenosis ≥ 50%; aortic arch atheroma ≥ 4 mm; intracranial artery stenosis ≥ 50% and presence of ischemic myocardial scar. The scar pattern was classified as ischemic if its distribution was sub-endocardial to transmural within a coronary vascular territory and if scar was associated with segmental systolic dysfunction on corresponding cine images. Atherosclerotic burden will be classified in 0, 1, 2, 3 and 4 atherosclerotic levels according to the number of arterial territories affected by at least one significant abnormality.
To assess the additional yield of cci-MR in cryptogenic patients and in those with embolic stroke of undetermined source (ESUS) with the reference strategy (ref Hart et al., Lancet Neurol. 2014:13:429-438.) | Within 8 days after hospitalization
  Etiology subtype according to ASCOD classification with the reference strategy + cci-MR in cryptogenic patients and in the subgroup of patients with ESUS with the reference strategy
To assess the rate of TEE recommended according to the opinion of the expert committee from data obtained with cci-MR and the reference strategy | Within 8 days after hospitalization
  Presence or absence of recommendation to realize a TEE according to the opinion of the expert committee from data obtained with cci-MR and with the reference strategy
To assess the rate of additional cardiologic advice recommended according to the opinion of the expert committee from data obtained with cci-MR and with the reference strategy | Within 8 days after hospitalization
  Presence or absence of recommendation to have a cardiologic advice according to the opinion of the expert committee from data obtained cci-MR and with the reference strategy
To assess the preventive treatment recommended (antithrombotic drugs and specific treatments) according to the opinion of the expert committee from data obtained with cci-MR and with the reference strategy | Within 8 days after hospitalization
  Presence or absence of recommendation of having antiplatelet, anticoagulant, and of having a specific care (carotid surgery, PFO closure…) according to the opinion of the expert committee from data obtained with cci-MR and with the reference strategy
To assess the feasibility of the examinations (rate of completed examinations, deadline to obtain each examination, deadline to obtain all examinations including in each strategy) | Within 8 days after hospitalization
  Presence or absence of full completed examinations, deadline between the date of ischemic stroke or TIA and each examination, deadline between the date of ischemic stroke or TIA and the end of all examinations including in each strategy
To assess the feeling of the patient about cci-MR and the reference strategy | Within 8 days after hospitalization
  Level of satisfaction of the patient about cci-MR and the reference strategy

CONTACTS AND LOCATIONS:
Overall Officials: MECHTOUFF Laura, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No